CLINICAL TRIAL: NCT02840461
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Multiple-Site Clinical Study to Evaluate the Therapeutic Equivalence and Safety of Ivermectin Cream 1% (Actavis Laboratories UT, Inc.) to SoolantraTM (Ivermectin) Cream 1% (Galderma) in the Treatment of Moderate to Severe Papulopustular Rosacea
Brief Title: Clinical Endpoint Study of Ivermectin 1% Cream
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 71591701
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Results first posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Moderate to Severe Papulopustular Rosacea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ivermectin Cream, 1% (Experimental): test product, manufactured by Actavis Laboratories UT, Inc.
  Interventions: Drug: Ivermectin Cream, 1%
- SoolantraTM (ivermectin) Cream, 1% (Active Comparator): reference product, manufactured by Galderma Laboratories, L.P.
  Interventions: Drug: Ivermectin Cream, 1%
- Placebo/Vehicle cream (Placebo Comparator): Placebo, manufactured by Actavis Laboratories UT, Inc.
  Interventions: Drug: Placebo/Vehicle cream

INTERVENTIONS:
Drug: Ivermectin Cream, 1%
  Arms: Ivermectin Cream, 1%; SoolantraTM (ivermectin) Cream, 1%
Drug: Placebo/Vehicle cream
  Arms: Placebo/Vehicle cream

SUMMARY:
A randomized, double-blind, placebo-controlled, parallel-design, multiple-site clinical study to evaluate the therapeutic equivalence and safety of ivermectin cream 1% (Actavis Laboratories UT, Inc.) to SoolantraTM (ivermectin) cream 1% (Galderma) in the treatment of moderate to severe papulopustular rosacea.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent that meets all criteria of current FDA regulations.
2. Healthy male or non-pregnant, non-lactating female greater than or equal to 8 years of age with a clinical diagnosis of moderate to severe papulopustular rosacea, defined as the presence of:

   A total of 8 to 50 combined papules/pustules on the face, AND At least moderate erythema, AND Telangiectasia
3. Patient has a baseline Investigator's Global Evaluation (IGE) score of 3 (moderate) or 4 (severe) for rosacea severity (See Appendix A).
4. Females of child bearing potential must not be pregnant or lactating at Screening (as confirmed by a negative urine pregnancy test with a sensitivity of less than 25 mlU/mL or equivalent units of human chorionic gonadotropin). Women of childbearing potential must agree to the use of a reliable method of contraception (e.g., total abstinence, IUD, a double-barrier method [such as condom plus diaphragm with spermicide], oral, transdermal, injected or implanted non- or hormonal contraceptive), throughout the study. If the female is using a hormonal contraceptive, the same product must be taken for 3 months prior to Visit 1 and must agree not to replace with some other hormonal contraceptives during the study. A sterile sexual partner is not considered an adequate form of birth control.

   All females will be considered to be of childbearing potential unless they: Are post-menopausal, defined as women who have been amenorrheic for at least 12 consecutive months, without other known or suspected primary cause.

   Have been sterilized surgically or who are otherwise proven sterile (i.e., total hysterectomy, or bilateral oophorectomy) with surgery at least 4 weeks before Screening. Tubal ligation will not be considered a surgically sterile method.

   Female patients of childbearing potential are defined as Women without prior hysterectomy of at least 4 weeks, or who have had any evidence of menses in the past 12 months.

   Females who have been amenorrhea for more than or equal to 12 months, but the amenorrhea is possibly due to other causes, including prior chemotherapy, anti-estrogens, or ovarian suppression.
5. Free from any systemic or dermatologic disorder that, in the opinion of the Investigator, will interfere with the study results or increase the risk of adverse events.
6. Willing to minimize external factors that might trigger rosacea flare-ups (e.g., extreme temperatures, aggressive astringents, known offending foods such as spicy foods and thermally hot foods and drinks, prolonged sun exposure, strong winds, alcoholic beverages, and emotional stress) within 24 hours before the Screening visit.
7. Of any skin type or race, provided the skin pigmentation allows accurate evaluation of papulopustular rosacea.
8. Willingness and capability to cooperate to the extent and degree required by the protocol.

Exclusion Criteria:

1. Females who are pregnant, lactating or planning to become pregnant during the study period.
2. Patient has mild facial rosacea (less than 8 inflammatory lesions on the face) or very severe rosacea (more than 50 inflammatory lesions).
3. Patient has mild erythema.
4. Patient has a baseline IGE score of 0, 1 or 2.
5. Patient has a skin condition on the face that would interfere with the diagnosis or assessment of rosacea (e.g., dermatitis, psoriasis, squamous cell carcinoma, eczema, acneform eruptions caused by medications, steroid acne, steroid folliculitis, bacterial folliculitis).
6. Patients with excessive facial hair, such as beards, sideburns, moustaches, etc., that would interfere with diagnosis or assessment of rosacea.
7. Patients with tattoos or excessive facial scarring that, in the Investigator's opinion, may interfere with the evaluation of the patient's rosacea.
8. Patients with active facial sunburn, peeling from sunburn, or patients that will be exposed to excessive sunlight during the study.
9. Patient has significant history or current evidence of chronic infectious disease, system disorder, organ disorder or other medical condition that in the Investigator's opinion would place the study patient at undue risk by participation.
10. Any patient (male or female) who has started, or changed hormonal therapy within 3 months of the baseline visit (this includes hormonal contraceptives). Patients who have been on stable hormone therapy for at least 3 months and whose therapy is considered unlikely to be changed for the duration of the study will be eligible.
11. History of hypersensitivity or allergy to study drug, or other ingredients of the formulation.
12. Use within 6 months prior to baseline of oral retinoids (e.g., Accutane) or therapeutic vitamin A supplements of greater than 10,000 units/day (multivitamins are allowed).
13. Use for less than 3 months prior to baseline of estrogen- and/or progestin-containing oral, injectable, implant, or transdermal contraceptives; use of such therapy must remain constant throughout the study.
14. Use within 1 month prior to baseline of 1) topical retinoids to the face, 2) systemic (e.g., oral or injectable) antibiotics known to have an impact on the severity of facial rosacea (e.g., containing tetracycline and its derivatives, erythromycin and its derivatives, sulfamethoxazole, or trimethoprim), 3) systemic steroids, 4) photodynamic therapy (including laser and other light therapies), or 6) cosmetic procedures (e.g., superficial chemical peels, exfoliation or microdermabrasion of the face).
15. Use within 2 weeks prior to baseline of 1) topical corticosteroids, 2) topical antibiotics, 3) topical anti-inflammatory agents or 4) topical medications for rosacea (e.g., metronidazole, azelaic acid, sodium sulfacetamide, ivermectin) 5) immunosuppressive drugs, 6) anticoagulant therapy.
16. Use of any other topical products applied to the target site.
17. Use of systemic corticosteroids. The use of inhaled corticosteroids up to less than 1mg per day is acceptable.
18. Use of antipruritics, including antihistamines, within 24 hours of study visits.
19. Patients who use make-up must have used the same brands/types for a minimum period of 14 days before study entry and must agree to not change brand or frequency of use throughout the study.
20. Presence of carcinoid, pheochromocytoma, or other causes of systemic flushing.
21. Presence of acne conglobata, acne fulminans, secondary acne or severe acne requiring systemic treatment.
22. Ocular rosacea (e.g., conjunctivitis, blepharitis, or keratitis) of sufficient severity to require topical or systemic antibiotics.
23. Receipt of any drug as part of a research study within 30 days before dosing.
24. Employees of the research center or Investigator.
25. Patients who are illiterate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Investigator site 1, Arlington Heights, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ivermectin Cream, 1%: Test product, manufactured by Actavis Laboratories UT, Inc.
  Ivermectin Cream, 1%
- SoolantraTM (Ivermectin) Cream, 1%: Reference product, manufactured by Galderma Laboratories, L.P.
  Ivermectin Cream, 1%
- Placebo/Vehicle Cream: Placebo, manufactured by Actavis Laboratories UT, Inc.
  Placebo/Vehicle cream
Period: Overall Study
Arm/Group | Ivermectin Cream, 1% | SoolantraTM (Ivermectin) Cream, 1% | Placebo/Vehicle Cream
Started | 259 | 257 | 114
Completed | 236 | 235 | 100
Not Completed | 23 | 22 | 14
Not completed — Adverse Event | 1 | 5 | 3
Not completed — Lost to Follow-up | 10 | 7 | 6
Not completed — Non-Comliance with Dosing Requirements | 0 | 1 | 0
Not completed — Protocol Violation | 2 | 3 | 1
Not completed — Withdrawal by Subject | 10 | 6 | 2
Not completed — Worsening of Symptom & Kit Error | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ivermectin Cream, 1% | SoolantraTM (Ivermectin) Cream, 1% | Placebo/Vehicle Cream | Total
Number analyzed (Participants) | 259 | 257 | 114 | 630
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (15.4) | 50.3 (15.0) | 51.1 (14.1) | 51.1 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 182 | 85 | 449
  Male | 77 | 75 | 29 | 181
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 136 | 133 | 65 | 334
  Not Hispanic or Latino | 123 | 124 | 49 | 296
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 2
  White | 253 | 253 | 114 | 620
  More than one race | 3 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 12 in the Number of Inflamed (Papules/Pustules) Lesions of Rosacea.
Description: Bioequivalence of the test to reference was considered to have been demonstrated if the 90% confidence interval for the test to reference ratio for the percent change from baseline to Week 12 in the number of inflamed lesion counts was within [80%, 125%].
Time Frame: Baseline and 12 Weeks
Population: Modified Intent-to-Treat Population
Measure: Least Squares Mean (Standard Error); unit: percentage of change from baseline
Groups:
- Vehicle Cream: Placebo cream (manufactured by Actavis Laboratories UT, Inc.)
Arm/Group | Ivermectin Cream, 1% | SoolantraTM (Ivermectin) Cream, 1% | Vehicle Cream
Number analyzed (Participants) | 251 | 248 | 111
percentage of change from baseline | -64.87 (2.03) | -64.87 (2.03) | -55.04 (2.92)
Statistical Analysis 1: Comparison: Ivermectin Cream, 1% vs SoolantraTM (Ivermectin) Cream, 1%; Test type: Equivalence — Therapeutic equivalence of the Test product to the Reference product based on the primary endpoint was evaluated in the PP population. If the confidence interval is within 80-125% for the primary endpoint, then the Test and Reference treatments are considered therapeutically equivalent; Mean Difference (Net) = 103.51, 90% CI 2-sided [97.95 to 110.00]
Statistical Analysis 2: Comparison: Ivermectin Cream, 1% vs Vehicle Cream; Test type: Superiority; p = 0.0027, ANOVA; Mean Difference (Net) = -9.83, 95% CI 2-sided [-16.24 to -3.42]
Statistical Analysis 3: Comparison: SoolantraTM (Ivermectin) Cream, 1% vs Vehicle Cream; Test type: Superiority; p = 0.0028, ANOVA; Mean Difference (Net) = -9.83, 95% CI 2-sided [-16.25 to -3.40]

2. Secondary Outcome: The Percentage of Patients With a Clinical Response of "Success".
Description: The secondary endpoint was the percentage of patients with a clinical response of "success" using the IGE at Week 12. At Visit 1, the IGE had to be 3 or 4 for the patient to be eligible for inclusion.
Time Frame: Baseline to Week 12
Population: Modified Intent-To-Treat Population
Measure: Count of Participants; unit: Participants
Groups:
- Vehicle Cream: Placebo Cream: manufactured by Actavis Laboratories UT., Inc.
Arm/Group | Ivermectin Cream, 1% | SoolantraTM (Ivermectin) Cream, 1% | Vehicle Cream
Number analyzed (Participants) | 251 | 248 | 111
Participants | 117 | 108 | 45
Statistical Analysis 1: Comparison: Ivermectin Cream, 1% vs SoolantraTM (Ivermectin) Cream, 1%; Test type: Equivalence — If the 90% confidence interval (with Yates correction) for the difference between the proportion of patients in the Test and Reference groups considered to be a clinical success was contained within the pre-defined equivalence limits [-20%, +20%], the therapeutic equivalence of the Test to Reference product was considered supported; Mean Difference (Net) = 5.8, 90% CI 2-sided [-2.7 to 14.2]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Ivermectin Cream, 1% | SoolantraTM (Ivermectin) Cream, 1% | Placebo/Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/259 | 0/257 | 0/114
Serious Adverse Events (participants affected / at risk) | 0/259 | 0/257 | 0/114
Other Adverse Events (participants affected / at risk) | 18/259 | 24/257 | 14/114
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivermectin Cream, 1% (N=259) | SoolantraTM (Ivermectin) Cream, 1% (N=257) | Placebo/Vehicle Cream (N=114)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Application site eczema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Application site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Application site pain (General disorders) | 2 (3) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pnuemonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (6) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes